CLINICAL TRIAL: NCT03010891
Title: Effects of Bundled Supportive Interventions on Preterm Infants' Stress-Related Outcomes
Brief Title: Effects of Bundled Supportive Interventions on Preterm Infants' Stress-Related Outcomes During Invasive Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hsiang-Yun Lan, Investigator, National Defense Medical Center, Taiwan, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2-104-05-157
Record Dates: First submitted 2016-12-29; First posted 2017-01-05 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Preterm Infants; Stress
Keywords: Preterm infant; Stress; Salivary DHEA; Salivary cortisol; Actigraphy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control condition (Active Comparator): Preterm infants in the control condition will receive only usual NICU care, plus positioning and gentle touch during intrusive procedures.
  Interventions: Behavioral: Usual NICU care
- experimental condition (Experimental): The bundle of supportive interventions will be designed to alleviate preterm infants' stress/pain from birth to discharge from the hospital NICU.
  Interventions: Behavioral: The bundle of supportive interventions

INTERVENTIONS:
Behavioral: The bundle of supportive interventions — usual NICU care +positioning + gentle touch + modulating infant states + facilitated tucking + NNS+ oral sucrose+ routine KMC > 45 minutes
  Arms: experimental condition
Behavioral: Usual NICU care — usual NICU care + positioning + gentle touch +routine KMC < 20 minutes
  Arms: control condition

SUMMARY:
The proposed 2-year study has two specific aims: (1) to examine the effects of a "bundle" of supportive interventions on preterm infants' stress (salivary cortisol and dehydroepiandrosterone [DHEA] levels and physiological signals of infant distress), sleep, and physical activity in the NICU, and (2) to explore the relationships among preterm infants' salivary cortisol and DHEA levels, physiological signals of infant distress, sleep, and physical activity. This randomized controlled trial will adopt a longitudinal repeated-measures design to examine the effects of bundled supportive interventions on preterm infants' stress (salivary cortisol and DHEA levels [using ELISA kit] and physiological signals of infant distress [using bedside electrocardiographic monitors]), sleep and physical activity (using ankle actigraphy) during their NICU hospitalization. Preterm infants (N=120) meeting the study criteria will be randomly assigned to one of two conditions: (1) control condition: usual NICU care + positioning + gentle touch +routine kangaroo mother care (KMC) < 20 minutes; (2) experimental condition: the bundle of supportive interventions (usual NICU care +positioning + gentle touch + modulating infant states + facilitated tucking + non-nutritive sucking + oral sucrose+ routine KMC > 45 minutes. Outcome variables will include infants' biological responses to stress (salivary cortisol, salivary DHEA, and physiological signals of infant distress), sleep patterns, and physical activity.

DETAILED DESCRIPTION:
Background and purpose: Preterm infants need to receive intensive care in a neonatal intensive care unit (NICU) to survive, but this care exposes them to painful procedures and a stressful environment. Repeated, painful/stressful stimuli can disturb infants' sleep, change their physiological indicators, and affect their developing brain and organs, possibly resulting in negative, long-lasting developmental consequences. Therefore, NICU clinicians caring for these vulnerable infants have two important goals: to provide early interventions to minimize preterm infants' stress/pain and to improve their sleep and physical activity. The proposed 2-year study has two specific aims: (1) to examine the effects of a "bundle" of supportive interventions on preterm infants' stress (salivary cortisol and dehydroepiandrosterone [DHEA] levels and physiological signals of infant distress), sleep, and physical activity in the NICU, and (2) to explore the relationships among preterm infants' salivary cortisol and DHEA levels, physiological signals of infant distress, sleep, and physical activity.

Methods: This randomized controlled trial will adopt a longitudinal repeated-measures design to examine the effects of bundled supportive interventions on preterm infants' stress (salivary cortisol and DHEA levels [using ELISA kit] and physiological signals of infant distress [using bedside electrocardiographic monitors]), sleep and physical activity (using ankle actigraphy) during their NICU hospitalization. Preterm infants (N=120) meeting the study criteria will be randomly assigned to one of two conditions: (1) control condition: usual NICU care + positioning + gentle touch +routine kangaroo mother care (KMC) < 20 minutes; (2) experimental condition: the bundle of supportive interventions (usual NICU care +positioning + gentle touch + modulating infant states + facilitated tucking + non-nutritive sucking + oral sucrose+ routine KMC > 45 minutes. Outcome variables will include infants' biological responses to stress (salivary cortisol, salivary DHEA, and physiological signals of infant distress), sleep patterns, and physical activity.

Expected outcomes: The study will fill a gap in knowledge about the effects of bundled supportive interventions on preterm infants' stress reactivity, sleep, and physical activity during hospitalization. This unique combination of physiological measurements of preterm infants' stress parameters and longitudinal design will provide results for establishing evidence-based clinical guidelines to provide atraumatic care to this population during intrusive procedures. Investigators also expect that bundling supportive interventions will minimize preterm infants' pain/stress as well as improve their sleep and physical activity. In the long term, the study results may help reduce the morbidity and complications due to preterm birth, save medical costs in neonatal care, and promote these infants' health and future developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* (1) gestational age (GA) > 28 weeks and < 37 weeks
* (2) birth weight < 2100g
* (3) stable condition (score < 22 on the Neonatal Therapeutic Intervention Scoring System [NTISS] for disease severity)
* (4) parents can speak, read and write Chinese
* (5) parents have no history of drug/alcohol abuse
* (6) parents agree to participate

Exclusion Criteria:

* (1) congenital anomalies
* (2) neurologic impairment including convulsion, intraventricular hemorrhage > grade II or periventricular leukomalacia
* (3) documented congenital or nosocomial (infection acquired at hospital after birth) sepsis
* (4) surgery
* (5) severe medical conditions requiring treatments such as cortisol supplementation, sedatives, muscle relaxants, antiepileptic, or analgesic drugs

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Preterm infant salivary cortisol | up to 3 months
  Accessed by salivary cortisol ELISA kit

SECONDARY OUTCOMES:
Preterm infant sleep | up to 3 months
  Accessed by Actigraphy
Preterm infant physiological signals of infant distress | up to 3 months
  Accessed by bedside electrocardiographic monitor
All preterm infants' physical activity are accessed by using Actigraphy | up to 3 months
  Accessed by Actigraphy
Preterm infant salivary DHEA levels | up to 3 months
  Accessed by salivary DHEA ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Jiuan Liaw, Professor, Study Chair — Professor, School of Nursing, 1National Defense Medical Center, Taipei, Taiwan, ROC.

IPD SHARING:
Plan to Share IPD: No